CLINICAL TRIAL: NCT00540462
Title: Prospective Randomized Trials of Gastric Bypass Surgery in Patients With Type II Diabetes Mellitus
Acronym: T2DM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Min-Sheng General Hospital (Other)
Responsible Party: Min-Sheng General Hospital, Min-Sheng General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Diabetes01
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-10

CONDITIONS: Type II Diabetes Mellitus
Keywords: Type II Diabetes Mellitus; Gastric bypass; Obese-related diabetes mellitus; Sugar control; treatment of obesity related diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): Medical Group
- 2 (Active Comparator): Surgical Group with gastric bypass
  Interventions: Procedure: gastric bypass
- 3 (Active Comparator): Sugical Group with Sleeve gastrectomy
  Interventions: Procedure: sleeve gastrectomy

INTERVENTIONS:
Procedure: gastric bypass
  Arms: 2
Procedure: sleeve gastrectomy
  Arms: 3

SUMMARY:
Although intensive medical treatment of diabetes has clearly been demonstrated to be worthwhile, it has not been a total success in diabetes treatment for a variety of reasons including lack of response to medication. Diabetes has been well demonstrated as a co-morbidity illness of obesity patients. In observation, with exclusion stomach and duodenum of bariatric surgery (gastric bypass), most morbidly obese patients (about 80%) with diabetes had a significant improved of sugar control. Base of this observation, we will try to find out the role surgical intervention (gastric bypass & sleeve gastrectomy) in obese-related diabetes.

DETAILED DESCRIPTION:
In observation, with exclusion stomach and duodenum of bariatric surgery (gastric bypass), most morbidly obese patients (about 80%) with diabetes had a significant improved of sugar control. Base on this observation, we will try to find out the role surgical intervention (gastric bypass and sleeve gastrectomy) in obese-related diabetes. With restriction of stomach volume and with or without duodenal exclusion, this randomized trials will find out the role of duodenal exclusion and the role of Ghrenin in obese-related type II DM patients. The initial observation of previous morbidly obese patients with type II DM, the DM seems a chronic disease which could be treated or controlled by surgical intervention, that's what we try to know more.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of T2DM for at least 6 months
* Mild to moderate obesity status(BMI 27 - 35 )
* Age : 30 - 60 year-old
* HbA1C > 8 %

Exclusion Criteria:

* With co-morbidity illness of cardiovascular system
* DM related nephropathy (Cre >2.0 mg/dl)
* Pulmonary embolism or uncontrolled coagulopathy in 6 months
* HBV or HCV hepatitis or liver cirrhosis, inflammatory colon disease, Cushing syndrome
* s/p organ transplantation
* Previously Bariatric surgery, gastrointestinal surgery, or abdominal sepsis
* Alcoholic or drug abuser
* Psychological disease.
* HIV or TB patient

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-08 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Measure sugar levels, HbA1c levels, and medication needed. OGTT, MGTT. | 1st, 2nd, 3rd, 4th, 5th, 6th, 9th, 12th months

SECONDARY OUTCOMES:
Comparing the DM controls between Medical and Surgical treatment In surgery groups, compare the bypass surgery and sleeve gastrectomy | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Lee WeiJei, M.D, Ph.D, Principal Investigator — MSGH
Locations (1):
- MinSheng Genral Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Lee WJ, Chong K, Ser KH, Lee YC, Chen SC, Chen JC, Tsai MH, Chuang LM. Gastric bypass vs sleeve gastrectomy for type 2 diabetes mellitus: a randomized controlled trial. Arch Surg. 2011 Feb;146(2):143-8. doi: 10.1001/archsurg.2010.326. PMID 21339423